CLINICAL TRIAL: NCT01718106
Title: Randomized Study to Evaluate Segmental Late Loss Comparing Two PCI Strategies Using a Long Stent vs 2 Shorter Stents to Treat Long or Tandem Coronary Stenosis.
Brief Title: Single Long vs Two Short Overlapping Bioabsorbable Polymer DES
Acronym: ROCCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, Dr Alessandro Lupi, Cardiologia Ospedaliera, AOU Maggiore della Carità, Novara., Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 846/CE
Record Dates: First submitted 2012-10-27; First posted 2012-10-31 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; drug eluting stent; bioabsorbable polymer; percutaneous coronary intervention; restenosis; late thrombosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single long bioabsorbable polymer DES (Active Comparator): Patients with long coronary stenosis treated by a single long bioabsorbable polymer DES
  Interventions: Device: implantation of a bioabsorbable polymer DES
- Two bioabsorbable polymer DES in overlapping (Active Comparator): patients with long coronary artery stenosis tretaed by 2 bioabsorbable polymer DES with minimal overlapping
  Interventions: Device: implantation of a bioabsorbable polymer DES

INTERVENTIONS:
Device: implantation of a bioabsorbable polymer DES — implantation in patients with long coronary artery stenosis of a single long or two shorter overlapped bioabsorbable polymer DES

SUMMARY:
Multiple overlapping drug-eluting coronary stents (DES) are usually needed to treat long coronary stenoses but this strategy is expensive and the response to overlapping DES has not been extensively studied. The recent availability of bioabsorbable polymer DES could allow treatment of long coronary stenoses without leaving gross burden of non-absorbable polymer in the vessel wall, even in case of overlapping stents.

Thus we planned to evaluate which of the 2 strategies, namely using a single long biabsorbable DES or two shorter biabsorbable DES with minimal overlapping, is better in treating long coronary stenoses.

The study is a spontanous randomized multicenter open-label study. A maximum of 300 patients with stable angina and at leat 1 coronary stenosis >28mm and <40mm of length will be randomized in 1:1 fashion by a Web-based electronic CRF. The long stent group (Group A) will be treated by a single 44mm Biomime DES (II generation DES with bioabsorbable polymer, Meril Life Sciences Pvt. Ltd., Gujarat, India). The short stent group (Group B) will be treated by 2 short Biomime DES positioned with minimal overlapping. The primary end-point of the study will be the 6 moth in-stent late lumen loss. Seconadry end-points will be 1, 6 and 12 month overall mortality, myocardial infarction, target vessel revascularization, stent thrombosis and MACE (combination of the 3 previous clinical end-points). Patients will be evaluated by 6-month control coronary angiography and late lumen loss in the stented vessel will be measured in a quantitative coronary angiography Core Lab (Cardioimaging Centre, Novara, Italy)

ELIGIBILITY:
Inclusion Criteria:

1. De novo coronary artery stenosis in a major coronary artery branch (reference diameter 2.5-4.0 mm) with a lenght >28mm and <39mm
2. Symptoms or instrumental evidence of myocardial ischemia:

   * Chronic stable angina [Canadian Cardiovascular Society Classification]
   * Unstable angina with ECG changes or troponin release (Braunwald Class IB-C, IIB-C, or IIIB-C)
   * Stress ECG or myocardial perfusion imaging or stress echocardiography positive for inducible myocardial ischemia
3. Written informed consent to the study

Exclusion Criteria:

1. Pregnancy or lactation
2. Acute ST elevation myocardial infarction (primary angioplasty)
3. Cardiogenic shock
4. Known allergic reactions to aspirin, clopidogrel, prasugrel, heparin, enoxaparin, bivalirudin, steel, chromium, iodiate contrast medium
5. Platelets <75.000/mm3 or >700.000/mm3 or white blood cells <3.000/mm3.
6. Partecipation to other studies.
7. Active or <3 months peptic ulcer or gastrointestinal bleeding
8. Planned major surgery non delayable .
9. Comorbidities limiting life expectancy to <1 year.
10. Unprotected left main disease as target lesion
11. Chronic total occlusion as target lesion
12. Bifurcation with side branch > 2.5mm as target lesion
13. Restenosis as target lesion
14. saphenous vein graft as target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
follow up in-stent late lumen loss | 6-month
  difference between the in-stent coronary lumen measure obtained immediately after coronary percutaneous intervention and the in-stent coronary lumen measure at follow up

SECONDARY OUTCOMES:
overall mortality | 1 year
  mortality for all causes
Myocardial infarction | 1 year
  Myocardial infarction (universal definition of myocardial infarction, ACC/AHA/ESC statement) in the territory of the treated coronary artery
target vessel revascularization | 1 year
  revascularization of the treated coronary vessel by repeated percutaneous coronary intervention or coronary artery bypass grafting due to restenosis and or symptoms or instrumental signs of myocardial ischemia
Stent thrombosis | 2 years
  Coronary stent thrombosis according to ARC definition
MACE (major coronary adverse event) | 1 year
  combined endpoint = presence of overall death or myocardial infarction or target vessel revascularization or stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, MD, Principal Investigator — AOU Maggiore della Carità - Novara; Angelo S Bongo, MD, Study Chair — AOU Maggiore della Carità - Novara
Locations (1):
- Ospedale Maggiore della Carità, Novara, Italy